CLINICAL TRIAL: NCT00734227
Title: TIPS Versus Portacaval Shunt for Acute Bleeding Varices in Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Marshall J. Orloff, M.D., University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TvSSTUDY
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-07

CONDITIONS: Bleeding
Keywords: Survival and control of hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Randomization: By the blind card method to TIPS or emergency portacaval shunt. Diagnostic Workup: Completed within 6hr. Rapidity of Therapy: Within 24 hr. Failure of Therapy: Bleeding requiring >6u PRBC in first 7 days, or 8 units PRBC during 12 months.
  Rescue Crossover Therapy: When primary therapy has failed. Followup: Lifelong data collection on line, analysis by biostatistician Florin Vaida, PhD. External Advisory, Data Monitoring and Safety Committee by 3 senior academicians.
  Procedure: Emergency portacaval shunt.
  Interventions: Procedure: Emergency portacaval shunt
- B (Active Comparator): Procedure: Emergency TIPS.
  Interventions: Other: Emergency TIPS

INTERVENTIONS:
Procedure: Emergency portacaval shunt
  Arms: A
Other: Emergency TIPS
  Arms: B

SUMMARY:
In unselected cirrhotic patients with acute portal hypertension-related bleeding to compare the effectiveness in control of bleeding, mortality rate, duration of life, quality of life, and economic costs of two widely used treatment measures: (1) emergency transjugular intrahepatic portal-systemic shunt (TIPS), and (2) emergency portacaval shunt.

ELIGIBILITY:
Inclusion Criteria:

* All patients with UGI bleeding who are shown to have the findings of cirrhosis and esophagogastric varices or portal hypertensive gastropathy and require 2 or more units of blood transfusion will be included.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 1996-07; Primary Completion 2003-10 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Survival | 10 years

SECONDARY OUTCOMES:
Control of bleeding and quality of life | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Marshall J. Orloff, M.D., Principal Investigator — UCSD Medical Center
Locations (1):
- UCSD Medical Center, San Diego, California, United States

REFERENCES:
- [Derived] Orloff MJ. Fifty-three years' experience with randomized clinical trials of emergency portacaval shunt for bleeding esophageal varices in Cirrhosis: 1958-2011. JAMA Surg. 2014 Feb;149(2):155-69. doi: 10.1001/jamasurg.2013.4045. PMID 24402314
- [Derived] Orloff MJ, Vaida F, Haynes KS, Hye RJ, Isenberg JI, Jinich-Brook H. Randomized controlled trial of emergency transjugular intrahepatic portosystemic shunt versus emergency portacaval shunt treatment of acute bleeding esophageal varices in cirrhosis. J Gastrointest Surg. 2012 Nov;16(11):2094-111. doi: 10.1007/s11605-012-2003-6. Epub 2012 Sep 25. PMID 23007280